CLINICAL TRIAL: NCT03562091
Title: Observational Study on Perception of Information and Quality of Life in Neuroendocrine Tumor on Lanreotide Autogel
Brief Title: Perception of Information and Quality of Life in Neuroendocrine Tumour on Lanreotide Autogel
Acronym: OPERA
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-FR-52030-371
Record Dates: First submitted 2018-05-17; First posted 2018-06-19 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — The study is an observational evaluation that does not affect physician practices, the physician-patient relationship, or the care of subjects. The prescriptions will be decided prior to inclusion of the subject into the study. The information will be recorded using the data available in the medical file or collected during the visit (as part of the routine subject management).

SUMMARY:
The purpose of the study is to evaluate, in standard practice, the change in information received and perceived by the patient, extension of the disease and its treatment. These parameters will be evaluated by means of validated self-administered questionnaires that can be used in standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Gastroenteropancreatic neuroendocrine tumor (GEPNET), histologically proven, grade

  1 or 2,
* Subject eligible for antitumor treatment initiation with lanreotide autogel*, alone or combined with other therapies, selected freely and prior to inclusion in the study by the physician,
* Subject able to complete a self-administered evaluation questionnaire during initiation visit and liable to be seen again within 6 months of the initial visit based on the physician's usual practices
* Having consented in writing to his/her data being accessed for participation in the study.

Exclusion Criteria:

* Previously treated by lanreotide autogel
* Simultaneously participating in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Gastroenteropancreatic neuroendocrine tumor (GEPNET) from Primary care clinics
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Absolute variation on the score (standardized on a scale from 0 to 100) of the 3 targeted dimensions (disease, treatments and supportive care) of the self-administered Quality of Life Questionnaire (QLQ) QLQINFO25 | Change from Baseline to Month 6

SECONDARY OUTCOMES:
Change from baseline to Month 3 of the 3 targeted dimensions (disease, treatments and supportive care (ie, other services)) of QLQ-INFO25 self-administered questionnaire | Change from Baseline to Month 3
Changes from baseline to Month 3 and Month 6 on dimensions of the QLQ-INFO25 self-administered questionnaire not part of the primary endpoint | Change from Baseline to Month 3 and 6
Change from baseline to Month 3 and Month 6 in quality of life using QLQ-C30 questionnaire | Change from Baseline to Month 3 and Month 6
Changes of symptoms assessments (presence of symptoms or not) as part of the monitoring of the Neuroendocrine Tumor (NET) | Change from Baseline to Month 3 and to Month 6
Changes of biochemical markers expressed in terms of results (decrease, stable, increase) as part of the monitoring of the NET | Change from Baseline to Month 3 and to Month 6
Progression (yes/no) of NET on imaging as part of the monitoring of the NET | Month 3 and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen Central Contact, Paris, France